CLINICAL TRIAL: NCT00108342
Title: Nicotine Delivery Systems: Research and Treatment
Brief Title: Nicotine Delivery Systems: Research & Treatment
Acronym: NDS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Common comorbidities of Veterans precluded sufficient recruitment and enrollment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NEUA-015-07S; NCT00876239 (obsolete NCT alias)
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Smoking
Keywords: nicotine; drug therapy; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Chewing Gum; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine Replacement Treatment (NRT) Sampling (Active Comparator): Sampling = 3 minute testing of each of 6 NRTs (3 forms x 2 dosages)
  2 mg and 4 mg nicotine gum; 2 mg and 4 mg nicotine lozenges; frequent and infrequent puffing on a nicotine inhaler (can yield 4 mg from 10 mg device).
  Interventions: Drug: Nicotine gum - 2 mg and 4 mg; Drug: Nicotine lozenges - 2 mg and 4 mg; Drug: Nicotine inhaler (4 mg yield) - low and high "dosage" by frequency of puffing
- NRT Computer Learning (Sham Comparator): Computer learning: learning about 6 NRTs (3 forms x 2 dosages) by computer only
  Interventions: Other: Computer learning

INTERVENTIONS:
Drug: Nicotine gum - 2 mg and 4 mg
  Other Names: Nicorette gum
  Arms: Nicotine Replacement Treatment (NRT) Sampling
Drug: Nicotine lozenges - 2 mg and 4 mg
  Other Names: Nicorette Commit lozenges
  Arms: Nicotine Replacement Treatment (NRT) Sampling
Drug: Nicotine inhaler (4 mg yield) - low and high "dosage" by frequency of puffing — can yield 4 mg from 10 mg device - infrequent and frequent puffing
  Other Names: Nicotrol
  Arms: Nicotine Replacement Treatment (NRT) Sampling
Other: Computer learning
  Arms: NRT Computer Learning

SUMMARY:
The purpose of this study is to determine whether sampling nicotine replacement treatments (NRTs) is superior to learning about them by computer. Testing also covers preferences among the treatments. Subjects will be enrolled veterans who smoke.

Hypothesis: Direct experience ("sampling") of NRTs will increase knowledge about NRTs, motivation/confidence, use of NRTs and quit attempts in contrast to learning about NRTs by computer.

DETAILED DESCRIPTION:
The study was designed to compare sampling of several nicotine replacement treatments (NRTs) in contrast to a computer learning control. The NRTs include: 2 dosages of nicotine gum, 2 dosages of nicotine lozenges and 2 dosages of oral nicotine inhalers. In the sampling group, each participant tries each of the 6 NRTs for 3 minutes. In the control, the individuals read about the treatments. Dependent measures include: quit attempts, use of NRTs, preferences among NRTs, and learning and motivation.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled veteran who smokes.

Exclusion Criteria:

* Any event or condition that could be exacerbated by the local effects of nicotine treatments (e.g., throat or stomach problems; any kind of wheezing from a condition or medication)
* other criteria as determined by PI and study physicians
* reactions to menthol (inhaler) or to aspartame (lozenge)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina G. Schneider, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 enrollees gave their signed consent and were then screened for participation; a total of 17 participated in testing.
Groups:
- NRT Sampling: Sampling = actual 3 minute testing of each of 6 NRTs (3 forms x 2 dosages)
  Nicotine gum - 2 mg and 4 mg
  Nicotine lozenges - 2 mg and 4 mg
  Nicotine inhaler - infrequent and frequent puffing for dosage (can yield 4 mg from 10 mg device)
Period: Overall Study
Arm/Group | NRT Sampling | NRT Computer Learning
Started | 8 | 9
Completed | 7 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NRT Sampling | NRT Computer Learning | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Quit Attempts, Use of NRTs, Preference Among NRTs
Description: In addition to quit attempts, use of NRTs, and preference among NRTs, we also planned to assess learning and changes in motivation at all visits. Unfortunately, the study was terminated due to common comorbidities among the Veterans that precluded entry into the study. Due to the consequent small sample size, we did not analyze any data.
Time Frame: At testing, at follow-up
Population: The study was terminated and the data were not analyzed due to the small sample size.
Arm/Group | NRT Sampling | NRT Computer Learning
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Assessment of adverse events was carried out by the PI, a Study Physician, and a Research Assistant. In this study, a non-serious adverse event was one that involved expected side effects of the medications. These were monitored for the NRT Sampling Arm during testing. Side effects were not assessed for the Computer Learning intervention.
Arm/Group | NRT Sampling | NRT Computer Learning
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 3/8 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRT Sampling (N=8) | NRT Computer Learning (N=0)
Nausea or Light-Headedness (Gastrointestinal disorders) | 3 (3) | 0 (0) — Side effects, for the non-serious events (light-headedness, nausea) were anticipated events and resolved quickly.

LIMITATIONS AND CAVEATS:
Limitations of the study: early termination of the study occurred due to widespread comorbidities precluding recruitment and enrollment of Veterans in this NRT trial. Specifically, the sample size was too small for any data analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No